CLINICAL TRIAL: NCT03046823
Title: Imaging-based Diagnosis of Diffuse Coronary Artery Disease and Quantification of Cardiac Remodeling in Obesity
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/501/C
Record Dates: First submitted 2016-05-31; First posted 2017-02-08 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen for future research
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to:

1. Characterize coronary artery disease (CAD) using CT Angiography (CTA) and scaling power law in 100 patients with obesity
2. Characterize cardiac remodeling using curvedness-based MRI in 100 patients with obesity
3. Compare the differences of cardiac and vascular remodeling in patients with metabolic syndrome and those without

DETAILED DESCRIPTION:
Background and Objectives:

Obesity is a common [affecting about 33% in the general adult population in US] metabolic disorder and it is increasing in prevalence in Singapore (about 10% of general adult population). As obesity is associated with cardiovascular disease (i.e., diffused coronary artery disease, DCAD) and leads to heart remodeling and heart failure, timely and accurate diagnosis of diffused coronary artery disease and its related cardiac remodeling in obesity is clinically urgently needed and this study aims to:

1. Characterize coronary artery disease (CAD) using CTA and scaling power law in 100 patients with obesity
2. Characterize cardiac remodeling using curvedness-based MRI in 100 patients with obesity
3. Compare the differences of cardiac and vascular remodeling in patients with metabolic syndrome and those without

Methodologies: 100 patients with obesity will be recruited for this study. All recruited patients will undergo fasting blood test for diagnosing metabolic syndrome. After that, they will undergo CTA and MRI within 1-2 weeks in-between. Patients' CTA images will be segmented and transformed to build 3D coronary artery models. The application of novel scaling power laws on these models will be used to diagnose diffuse CAD. Based on patients MRI images, the cardiac remodeling will be assessed with a novel curvedness-based imaging analysis method. The differences of cardiac and vascular remodeling in patients with metabolic syndrome and those without will be compared and analyzed.

In addition, subjects shall undergo ultrasound examination of the heart (echocardiogram), carotids and forearm arteries. Doppler and tissue-Doppler echocardiography constitutes the gold standard for cardiac diastolic function assessment. The findings shall be correlated with diastolic cine MRI findings. Carotid and forearm artery ultrasound allows investigation of vessel distensibility, carotid intimal thickness, pulse wave velocity, central arterial blood pressure estimation as well as endothelial function (via flow-mediated dilation). Perturbations of these parameters may be correlated with functional abnormalities on cardiac MRI and coronary disease on CT.

Subjects shall undergo fasting blood tests for metabolic profiling. The tests include blood levels of creatinine, electrolytes, insulin, glycated haemoglobin, fasting lipids, fasting sugar and postprandial sugar (75 g standard oral glucose load). Additionally blood samples shall be stored for potential future studies.

Clinical Significance: If success, this study in obesity should advance understanding of obesity-related CAD and cardiac and vessel remodeling, and further translate into improved diagnosis and treatment in obese patients.

Clinical Significance: If success, this study in obesity should advance understanding of obesity-related CAD and cardiac remodeling, and further translate into improved diagnosis and treatment in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-80.
2. with obesity BMI ≥27 .
3. Written informed consent obtained

Exclusion Criteria:

1. Individuals unable to provide informed consent.
2. Non-cardiac illness with life expectancy <2 years.
3. Pregnant state.
4. Allergy to iodinated contrast.
5. Significant arrhythmia; heart rate ≥ 100 beats/min; systolic blood pressure ≤90 mmHg.
6. Renal dysfunction (Glomerular filtration rate (GFR) <45 mL/min/1.73m2).
7. Contraindication to beta blockers or nitroglycerin.
8. Canadian Cardiovascular Society class IV angina.
9. with Cardiac pacemaker
10. with brain aneurysm or clips
11. with Electronic implants or prosthesis
12. with Eye metal foreign body injury
13. Severe claustrophobia
14. Thyroid dysfunction

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total recruitment number: 100 Participants' age limit of 21 to 80.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03-31 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of diffuse coronary artery disease using imaging techniques and quantification of cardiac remodeling in obesity | 36 months
  Imaging-based techniques used are MRI, CTA and Echocardiogram. Fasting blood tests will be carried out to determine metabolic syndrome. Cardiac and vascular remodeling in participants with metabolic syndrome and those without will be compared and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: RU SAN TAN, Principal Investigator — National Heart Centre
Locations (1):
- National Heart Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided